CLINICAL TRIAL: NCT06976138
Title: Sleep TO Prevent Post-surgical Pain
Acronym: STOPPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00454253; 1R01AG085712-01 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthristis
Keywords: total knee arthroplasty; knee replacement; koa; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Cognitive Behavioral Therapy; Sleep

STUDY DESIGN:
Intervention Model Description: randomized controlled, 3-parallel arm, trial
Who Masked: Participant
Masking Description: Only the interventionist and biostatistician will have access to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy + Morning Bright Light exposure (Experimental): Cognitive-Behavioral Therapy for Insomnia. This program will focus on changing the participant's sleep patterns, activities, and habits.
  Morning Bright Light involves wearing glasses (Re-Timer Device) that give off a special type of bright light for one full hour in the morning. The participant will be asked to wear these glasses every morning for about four weeks before surgery, four weeks after surgery and again for 1-week , 3-months after surgery. The participant will fill out a log to note light on/off times, any interruptions to light treatment, and primary activity while receiving the light exposure. The participant will also receive daily reminders to charge the device and turn it on during the scheduled time.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia; Device: Bright Light therapy via the Re-Timer®
- Cognitive Behavioral Therapy for Insomnia + Negative Ion exposure (Active Comparator): Cognitive-Behavioral Therapy for Insomnia. This program will focus on changing the participant's sleep patterns, activities, and habits.
  Negative Ion exposure. This procedure involves wearing a light weight negative ionizer (IonMi Device) around the neck for one hour in the morning. An ionizer gives off special negatively charged ions into the air. the participant will be asked to wear the device every morning for about four weeks before surgery, four weeks after surgery and again for 1-week, 3-months after surgery The participant will also receive daily reminders to charge the device and turn it on during the scheduled time.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia; Device: Negative Ion exposure via IonMi Device
- Sleep / Knee Osteoarthritis Education + Negative Ion exposure (Active Comparator): Sleep / Knee Osteoarthritis Education. This program will focus on increasing the participant's knowledge about sleep, sleep disorders and knee osteoarthritis.
  Negative Ion exposure. This procedure involves wearing a light weight negative ionizer (IonMi Device) around the neck for one hour in the morning. An ionizer gives off special negatively charged ions into the air. The participant will be asked to wear the device every morning for about four weeks before surgery, four weeks after surgery and again for 1-week, 3-months after surgery The participant will also receive daily reminders to charge the device and turn it on during the scheduled time.
  Interventions: Device: Negative Ion exposure via IonMi Device; Behavioral: Sleep / Knee Osteoarthritis Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Insomnia — This program will focus on changing the participant's sleep patterns, activities, and habits.
  Arms: Cognitive Behavioral Therapy + Morning Bright Light exposure; Cognitive Behavioral Therapy for Insomnia + Negative Ion exposure
Device: Bright Light therapy via the Re-Timer® — Subjects will conduct light treatment in the mornings at home for one hour using Re-timer® The participant will be asked to wear the device every morning for about four weeks before surgery, four weeks after surgery and again for 1-week, 3-months after surgery
  Arms: Cognitive Behavioral Therapy + Morning Bright Light exposure
Device: Negative Ion exposure via IonMi Device — This procedure involves wearing a light weight negative ionizer (IonMi Device) around neck for one hour in the morning. An ionizer gives off special negatively charged ions into the air. The participant will be asked to wear the device every morning for about four weeks before surgery, four weeks after surgery and again for 1-week, 3-months after surgery
  Arms: Cognitive Behavioral Therapy for Insomnia + Negative Ion exposure; Sleep / Knee Osteoarthritis Education + Negative Ion exposure
Behavioral: Sleep / Knee Osteoarthritis Education — This program will focus on increasing The participant's knowledge about sleep, sleep disorders and knee osteoarthritis.
  Other Names: koa Education
  Arms: Sleep / Knee Osteoarthritis Education + Negative Ion exposure

SUMMARY:
This research study is being done to compare different methods of addressing sleep problems before total knee replacement surgery. These methods include Cognitive Behavioral Therapy and light exposure.

DETAILED DESCRIPTION:
This research is being done to evaluate whether combining Cognitive Behavioral Therapy for Insomnia (talk therapy for insomnia) with Morning Bright Light exposure is more effective than Morning Negative Ion exposure combined with either Cognitive Behavioral Therapy for Insomnia or Sleep / Knee Osteoarthritis Education to reduce pain following total knee replacement surgery. This knowledge is needed to develop better ways to manage pain after surgery. Sleep problems are often not treated before or after surgery, so this may differ from the typical care received by adding a focus on sleep. People with knee osteoarthritis, who are 60 years old and older, who are scheduled to have unilateral (one knee) total knee replacement surgery for osteoarthritis and who have trouble falling or staying asleep, may join this study.

There are two possible devices that are being compared in this study.

* If the participants are in the Morning Bright Light exposure group, the participants will use the Re-timer®, a wearable bright light exposure device. This device is commercially available and in use by the general population. This device meets international ultraviolet and blue light hazard safety standards. The light intensities used in this study are greater than most indoor light, but much dimmer than sunlight on a bright day.
* If the participants are in the Negative Ionizer exposure group, the participants will use the IonPacific,"ionMi,"a wearable negative ionizer. This device is also commercially available and in use by the general population.

There have been reports of improved sleep and daytime symptoms associated with poor sleep for both Morning Bright Light and Negative Ionizer exposures. The use of Re-timer and IonMi in this research study is investigational. The word "investigational" means that the Re-timer and IonMi are not approved for marketing by the Food and Drug Administration (FDA).

Participation includes:

A virtual and in person screening and training visit 4, 1-hour long telehealth sessions scheduled each week before surgery 2, 30-minute telehealth sessions, 2-weeks after surgery and 3-months after surgery

This study will be using "blinding" which means only a few members of the study team will know what group / sleep program the participants have been assigned to until the study ends. In case of an emergency, the study doctor can quickly find out which sleep health program the participants have been assigned to receive.

During parts of the study, the device the participants are using may be deactivated in order to test the effects of an active study device compared to a deactivated device. At the end of the study, the team can provide information about the timing of device deactivation.

The participants will not be asked to change the clinical care currently being received for knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* People with knee osteoarthritis,
* 60 years old and older,
* scheduled to have unilateral (one knee) total knee replacement surgery for osteoarthritis and
* have trouble falling or staying asleep

Exclusion Criteria:

* currently using medications to help sleep
* have completed Cognitive Behavioral Therapy for Insomnia
* used either Bright Light or Negative Ion exposures in the past year
* have an inflammatory rheumatologic disorder, seizure disorder
* serious mental health disorder, Bipolar I disorder, substance or alcohol use disorder
* serious sleep or circadian rhythm disorder, untreated sleep apnea
* are pregnant or lactating
* have retinal pathology
* history of eye surgery (Lasik or cataract okay if more than 3 months ago)
* are taking disease-modifying antirheumatic drugs
* taking photosensitizing medications
* are unwilling to discontinue over the counter sleep aids (for example, melatonin) for at least 2 weeks before enrolling

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Chronic postsurgical pain as assessed by the Western Ontario and McMaster Universities Osteoarthritis Index | 3 and 6 months post-surgery
  Higher scores indicate higher pain. Asked to rate pain in different situations from 0 (no pain) to 10 (extreme pain) on Visual Analog Scale.

SECONDARY OUTCOMES:
Post-surgical pain as assessed by the Western Ontario and McMaster Universities Osteoarthritis Index Pain Severity | immediately post surgery, 6 weeks post surgery
  Higher scores indicate higher pain. Asked to rate pain in different situations from 0 (no pain) to 10 (extreme pain) on Visual Analog Scale.
Number of participants with Post-surgical opioid use | 6-weeks post-surgery, 3 and 6 months post surgery
  Opioid use after surgery reported in 7-day virtual diaries. Higher amounts mean higher intake of opioids. Participants will be asked to report prescribed opioids, how often being taken, and provide information via virtual pill count.
Insomnia Severity as assessed by the Insomnia Severity Index | pre-surgery, post-surgery 6-weeks, post surgery 3 months and 6-months
  Minimum score possible is 0, highest score 28. Higher scores indicate higher insomnia symptoms
Circadian Rest Activity Rhythm (RAR) assessed by actigraphy | pre-surgery, post-surgery 6-weeks, post surgery 3 months and 6-months
  Motion data from actigraphy monitors will be used to estimate circadian rest activities within and across 24-hour intervals. The investigators will model standard circadian RAR parameters derived from actigraphy data using both an extended cosinor analysis as well as non-parametric methods. For example, Pseudo F-statistics, and index of circadian rest activity rhythm, will be derived, and lower Pseudo F-statistics are related to less robust rest activity rhythm strength
Depressed mood as assessed by the Patient Health Questionnaire (PHQ-9) | pre-surgery, post-surgery 6-weeks, post surgery 3 months and 6 months
  Score range of 0-27. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.

OTHER OUTCOMES:
Post-surgical Physical Functioning as assessed by the Western Ontario and McMaster Universities Osteoarthritis Index Physical Functioning | 3 and 6 months post-surgery
  Higher scores indicate greater issues with physical functioning. Asked to rate difficulty performing different tasks from 0 (no difficulty) to 10 (extreme difficulty). Score range 0-68.
Wake After Sleep Onset Time (minutes) as assessed by actigraphy | pre-surgery, post-surgery 6-weeks, post surgery 3 months and 6 months
  Motion information from actigraphy monitors will be used with sleep diaries to provide information about sleep continuity patterns. This measure will use 1-week averages to determine wake after sleep time.
Total Sleep Time (minutes) as assessed by actigraphy | pre-surgery, post-surgery 6-weeks, post surgery 3 months and 6 months
  Motion information from actigraphy monitors will be used with sleep diaries to provide information about sleep continuity patterns. This measure will use 1-week averages to determine total sleep time.
Sleep Onset Latency (minutes) as assessed by actigraphy | pre-surgery, post-surgery 6-weeks, post surgery 3 months and 6 months
  Motion information from actigraphy monitors will be used with sleep diaries to provide information about sleep continuity patterns. This measure will use 1-week averages to determine sleep onset latency.
Sleep Efficiency as assessed by actigraphy | pre-surgery, post-surgery 6-weeks, post surgery 3 months and 6 months
  Motion information from actigraphy monitors will be used with sleep diaries to provide information about sleep continuity patterns. This measure will use 1-week averages to determine sleep efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Smith, PhD, Principal Investigator — Johns Hopkins University; Helen Burgess, PhD, Principal Investigator — University of Michigan; Robert R Edwards, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Mass General Brigham, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Final de-identified, anonymized data sets underlying all publications resulting from the proposed research involving human subjects will be shared with legitimate academic researchers and other community members with a legitimate scientific interest in the research. Where practicable, sharing will take place under a written agreement between the principal investigators prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the data sets. Study documentation (e.g., study protocols) will be made accessible via clinicaltrials.gov and via communication with the principal investigators to facilitate interpretation of the scientific data. Codebooks, other study documentation and deidentified data will be made available on the National Institute on Aging (NIA) National Archive of Computerized Data on Aging data (NACDA) repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The research community will have access to the data when the award ends. De-identified data will be provided after the requesters sign a Letter of Agreement detailing the purpose of the sharing request, information about the requesters and the requesters affiliations, mechanisms by which the data will be kept secure, and access restricted to the study team. The agreements will also state the recipient will not attempt to identify any individual whose data are included and will not share the data with anyone outside of the research team. NACDA make data available via public-use files (which would require agreement to NACDA's Terms of Use) or via restricted-use files (which would require a signed Restricted Data Use Agreement between the requestor's institution and the Johns Hopkins University as well as an application to request access).
Access Criteria: Pll data sharing will follow the guidelines and rules of the NIH and Johns Hopkins University's Institutional Review Board (IRB). Deidentified data will be managed as indicated in the informed consent. The Informed Consent will notify participants that the data will be shared. De-identified data will be share to the extent indicated in the informed consent. Final curated, de-identified, anonymized data sets underlying publications resulting from the proposed research involving human subjects will be generated and will be shared only to the extent indicated in the informed consent. Requesters will sign a Letter of Agreement with the Johns Hopkins University detailing the requesters planned uses of the data and mechanisms by which the data will be kept secure, and access restricted to the requesters study team with appropriate credentials and training in data security. NACDA's application for restricted-use data will be followed.